CLINICAL TRIAL: NCT06981104
Title: A Randomized, Double-blind, Controlled Clinical Study on the Efficacy and Safety of 0.05% Cyclosporine Eye Drops in the Treatment of Mild to Moderate Dry Eye
Brief Title: Tear Film Stability and Improvement of Asthenopia: Efficacy Observation of 0.05% Cyclosporine in Dry Eye Patients With Short BUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-0146
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-11

CONDITIONS: Dry Eye Disease (DED); Asthenopia
MeSH Terms: conditions — Dry Eye Syndromes; Asthenopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.05% cyclosporine froup(Group C) (Experimental)
  Interventions: Drug: 0.05% cyclosporine eyedrops
- 0.1% sodium hyaluronate group（Group S） (Placebo Comparator)
  Interventions: Drug: 0.1% sodium hyaluronate eye drop

INTERVENTIONS:
Drug: 0.05% cyclosporine eyedrops — 0.05% cyclosporine, one drop each time, twice a day
  Arms: 0.05% cyclosporine froup(Group C)
Drug: 0.1% sodium hyaluronate eye drop — 0.1% sodium hyaluronate, one drop each time, three times a day
  Arms: 0.1% sodium hyaluronate group（Group S）

SUMMARY:
At present, research on cyclosporine mainly focuses on patients with moderate to severe dry eye. Based on the importance of the vicious cycle of inflammation in the pathogenesis of dry eye and the mechanism of cyclosporine, investigators believe that it may also have therapeutic effects in patients with mild to moderate dry eye, and may have certain advantages compared to traditional artificial tear therapy. In summary, this study intends to use a randomized, double-blind, parallel controlled trial to evaluate the therapeutic efficacy and safety of 0.05% cyclosporine eye drops in patients with mild to moderate dry eyes.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old (including 18 and 75 years old), male or female;
2. Meets the diagnostic criteria for dry eye syndrome in China (2020) and is mild dry eye 1) Dry Eye Questionnaire (OSDI) score ≥ 13 points; 2) BUT ≤ 10 seconds or Schirmer I ≤ 5mm/5 minutes 3) Corneal staining positive ≤ 5 points.
3. At least one of OSDI, BUT, and Schirmer I meets the moderate standard OSDI ≥ 23 points; BUT<5 seconds; Schirmer I < 5mm/5min
4. The subjects themselves signed an informed consent form and voluntarily participated in this study.

Exclusion Criteria:

1. Women who are breastfeeding or pregnant, or men and women of childbearing age who are unable to use effective contraceptive methods during the study period;
2. Those who need to wear contact lenses during treatment;
3. Acute inflammation, infection, allergy, and trauma of the eyes;
4. There are obvious scars or keratinization on the eyelid margin;
5. Have undergone eye or eyelid surgery within the 6 months prior to enrollment;
6. Diagnosed with facial nerve paralysis or ocular nerve paralysis within 6 months prior to enrollment;
7. Currently using lacrimal duct embolization (permanent lacrimal plug or treatment with lacrimal plug within 6 months);
8. I am currently taking medication that may affect dry eye syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Fluorescent tear film breakup time | 8weeks
high-frequency component（HFC） | 8weeks
  HFC represents a slight deformation of the lens in a state of relative modulation stillness, indicating tremors in the ciliary muscle
ASQ-17 | 8weeks
  Asthenopia Survey Questionnaire (ASQ)-17,ASQ-17 covers 7 items of eye symptoms, 6 items of visual symptoms and 4 items of systemic and psychological symptoms with a total score of 51 and an optimal cut-off threshold value of 12.5[1].
  [1]Lin N, Li XM, Yang MY, Tian L, Li ZH, Mao JL, Zhang JF, Chen J, Lyu F, Deng RZ. Development of a new 17-item Asthenopia Survey Questionnaire using Rasch analysis. Int J Ophthalmol. 2023 Nov 18;16(11):1867-1875. doi: 10.18240/ijo.2023.11.20. PMID: 38028524; PMCID: PMC10626358.

CONTACTS AND LOCATIONS:
Locations (1):
- 1 Xihu Avenue, Shangcheng District, Hangzhou, Zhejiang, China, Hangzhou, Zhejiang, China